CLINICAL TRIAL: NCT03623139
Title: Effects of Basic Carbohydrate Counting Versus Standard Outpatient Nutritional Education: A Randomized Controlled Trial Focusing on HbA1c and Glucose Variability in Patients With Type 2 Diabetes (The BCC Study)
Brief Title: Effects of Basic Carbohydrate Counting Versus Standard Outpatient Nutritional Education in Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Steno Diabetes Center Copenhagen (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Bettina Ewers, Head of nutrition, MSc, Steno Diabetes Center Copenhagen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-18014918
Record Dates: First submitted 2018-07-18; First posted 2018-08-09 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Type2 Diabetes; Diabetes Mellitus, Type 2; Glucose Metabolism Disorders
Keywords: carbohydrates; basic carbohydrate counting; diet; type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Glucose Metabolism Disorders | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard nutritional education (Active Comparator): Control group
  Interventions: Behavioral: Standard nutritional education
- BCC (Experimental): Education and training i basic carbohydrate counting (BCC) plus standard nutritional education
  Interventions: Behavioral: Basic carbohydrate counting

INTERVENTIONS:
Behavioral: Standard nutritional education — Routine dietary care consists of three individual consultations with a trained dietitian. The individual guidance will be in accordance with the dietary guidelines in type 2 diabetes.
  Other Names: Routine dietary care in type 2 diabetes
  Arms: Standard nutritional education
Behavioral: Basic carbohydrate counting — The BCC concept is a group-based program consisting of three group sessions delivered by trained dietitians.
  Other Names: Education in BCC in addition to standard dietary care
  Arms: BCC

SUMMARY:
The aim of the study is to examine the health benefits of adding a concept in basic carbohydrate counting (BCC) to the routine outpatient nutritional education for adult patients with type 2 diabetes.

The study hypothesis is that training and education in the BCC concept will improve glycaemic control either by reducing HbA1c or the average plasma glucose variability more than offering the routine dietary care as a stand-alone dietary treatment.

DETAILED DESCRIPTION:
The trial has a parallel-group design with a study duration of 48 weeks for each participant (a 6-month intervention period and a 6-month follow-up period). A total of 226 patients will be enrolled in the trial. Participants will be randomized to one of two arms: 1) Standard medical and dietary care (control group) or 2) Structured training and education in the BCC concept in addition to standard medical and dietary care.

The primary objective is to evaluate the six months effect of structured training and education in the BCC concept compared to standard dietary care on glycaemic control as assessed by HbA1c or MAGE (mean amplitude of glycaemic excursions).

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Diabetes duration; from >12 months
* HbA1c between 53 and 97 mmol/mol
* Diet or any glucose-lowering medication
* Provided voluntary written informed consent

Exclusion Criteria:

* Practicing carbohydrate counting, as judged by the investigator
* Participated in a BCC group program within the last two years
* Low daily intake of carbohydrates (defined as below 25 E% or 100 g/day), as judged by the investigator
* Use of open CGM
* Use of a Free Libre device
* Use of an automated bolus calculator for carbohydrate counting, as judged by the investigator
* Gastroparesis
* Pregnancy or breastfeeding, or plans of pregnancy within the study period
* Uncontrolled medical issues, as judged by the investigator
* Concomitant participation in other clinical studies
* Unable to understand the informed consent and the study procedures

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2018-09-28 (Actual); Primary Completion 2022-08-16 (Actual); Study Completion 2022-08-16 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c | Baseline, 6 months
  mmol/mol
Change in mean amplitude of glycaemic excursions (MAGE) | Baseline, 6 months
  mmol/l

SECONDARY OUTCOMES:
Change in HbA1c | 12 months
  mmol/mol
Change in body weight | Baseline, 6 months, 12 months
  kg
Change in low-density lipoprotein cholesterol (LDL-C) | Baseline, 6 months, 12 months
  mmol/l
Change in high-density cholesterol (HDL-C) | Baseline, 6 months, 12 months
  mmol/l
Change in total cholesterol (TC) | Baseline, 6 months, 12 months
  mmol/l
Change in free fatty acids (FFA) | Baseline, 6 months, 12 months
  mmol/l
Change in triglycerides (TG) | Baseline, 6 months, 12 months
  mmol/l
Change in diastolic blood pressure | Baseline, 6 months, 12 months
  mm Hg
Change in systolic blood pressure | Baseline, 6 months, 12 months
  mm Hg
Change in waist circumference | Baseline, 6 months, 12 months
  cm
Change in hip circumference | Baseline, 6 months, 12 months
  cm
Change in total fat free mass | Baseline, 6 months
  gram
Change in total fat mass | Baseline, 6 months
  gram
Change in time in range (3.9-10.0 mmol/l) | Baseline, 6 months
  percent (%)
Changes in time spent in hypoglycaemia (<3.9 mmol/l) | Baseline, 6 months
  percent (%)
Change time spent in hyperglycaemia (e.g. >11.1 mmol/l) | Baseline, 6 months
  percent (%)
Change in standard deviation of mean plasma glucose | Baseline, 6 months
  mmol/l
Change in mathematical literacy | Baseline, 6 months, 12 months
  total score or percent (%)
Change in carbohydrate estimation accuracy | Baseline, 6 months, 12 months
  total score or %
Change in diet-related quality of life | Baseline, 6 months, 12 months
  total score or percent (%)
Change in perceived competences in diabetes | Baseline, 6 months, 12 months
  total score or percent (%)
Change in degree of autonomy-supportive dietitian | Baseline, 6 months, 12 months
  total score or percent (%)
Change in total energy intake | Baseline, 6 months
  kJ/day
Change in dietary intake of carbohydrates | Baseline, 6 months
  gram/day or percent of total energy (E%)
Change in dietary intake of total fat | Baseline, 6 months
  gram/day or percent of total energy (E%)
Change in dietary intake of saturated fatty acids (SFA) | Baseline, 6 months
  gram/day or percent of total energy (E%)
Change in dietary intake of monounsaturated fatty acids (MUFA) | Baseline, 6 months
  gram/day or percent of total energy (E%)
Change in dietary intake of polyunsaturated fatty acids (PUFA) | Baseline, 6 months
  gram/day or percent of total energy (E%)
Change in dietary intake of protein | Baseline, 6 months
  gram/day or percent of total energy (E%)
Change in dietary intake of added sugar | Baseline, 6 months
  gram/day , % of total energy or %
Change in intake of dietary fibre | Baseline, 6 months
  gram/day or g/MJ

OTHER OUTCOMES:
Change in physical activity level | Baseline, 6 months, 12 months
  total score or percent (%)
Change in urinary biomarkers of carbohydrate intake | Baseline, 6 months
  percent (%)

CONTACTS AND LOCATIONS:
Overall Officials: Bettina Ewers, MSc, Principal Investigator — Steno Diabetes Center Copenhagen
Locations (1):
- Steno Diabetes Center Copenhagen, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ewers B, Bruun JM, Vilsboll T. Effects of basic carbohydrate counting versus standard outpatient nutritional education (The BCC Study): study protocol for a randomised, parallel open-label, intervention study focusing on HbA1c and glucose variability in patients with type 2 diabetes. BMJ Open. 2019 Nov 21;9(11):e032893. doi: 10.1136/bmjopen-2019-032893. PMID 31753900

DOCUMENTS (2):
  • Study Protocol (2019-08-08): https://cdn.clinicaltrials.gov/large-docs/39/NCT03623139/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-25): https://cdn.clinicaltrials.gov/large-docs/39/NCT03623139/SAP_001.pdf